CLINICAL TRIAL: NCT04663568
Title: Levonorgestrel-releasing Intrauterine System: A Emerging Tool for Conservative Treatment of Pain and Bleeding After Tubal Ligation
Brief Title: Levonorgestrel-releasing Intrauterine System and Tubal Ligation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No fund was obtained for buying the hormonal IUD
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNG_TS
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Tubal Ligation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levonorgestrel-releasing intrauterine system (Other)
  Interventions: Device: Levonorgestrel-releasing intrauterine system

INTERVENTIONS:
Device: Levonorgestrel-releasing intrauterine system — Levonorgestrel-releasing intrauterine system will be inserted during the menstrual cycle

SUMMARY:
Today tubal sterilization is a simple, safe, and cost-effective method of achieving long-term contraception. Sterilization is an ideal method of permanent contraception in developing countries where access to health care providers is limited. The percentage of women who use sterilization as a method of contraception rises from about 5% between 20 and 24 years of age to almost 50% for those between 40 and 44 years of age. The most widely touted and most significant health benefit of tubal sterilization appears to be a reduced risk of ovarian cancer.

Post-tubal ligation syndrome includes pain during intercourse, aching lower back, premenstrual tension syndrome, uterine hemorrhage, and absence of menstruation. The syndrome is caused by blood circulation problems in and around the Fallopian tubes and ovaries, pressure on nerves, and intrapelvic adhesion. Since the symptoms of this syndrome are mild, simple symptomatic treatment is sufficient in most cases. In some cases, however, hysterectomy may be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 30-40 year
* Woman subjected to tubal ligation
* Women 12 month postpartum
* Non lactating women
* Nomedical disorders

Exclusion Criteria:

* contraindication for Levonorgestrel-releasing Intrauterine System
* Women with any uterine or ovarian pathology
* women refuse to participate

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The level of pain from before to 6 months after levonorgestrel-releasing intrauterine system insertion | 6 months
  visual analogue scale from 0 (minimum value) to 10 (maximum value)

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided